CLINICAL TRIAL: NCT02887495
Title: The Scleroderma Biorepository and Pathogenesis Study (STOP Scleroderma)
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Victoria Shanmugam, MD, Professor, George Washington University
Other Study IDs: 051427
Record Dates: First submitted 2015-02-03; First posted 2016-09-02 (Estimated); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Scleroderma
Keywords: scleroderma; biorepository
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Scleroderma bioreposiTOry and Pathogenesis Study (STOP Scleroderma) will help researchers use clinical data and human biospecimens to investigate why scleroderma patients develop certain complications from their disease. Patients with confirmed scleroderma, raynauds or positive autoantibodies are invited to participate. This research may help us understand how to prevent and treat scleroderma and other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Able to give informed consent.
* Diagnosed with scleroderma or with positive autoantibodies

Exclusion Criteria:

* < 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with scleroderma, raynauds, or with positive autoantibodies
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-07; Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Modified Rodnan Skin Score | 10 years

SECONDARY OUTCOMES:
Medsger Severity Score | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Victoria K Shanmugam, MD, Principal Investigator — The George Washington University
Locations (1):
- Victoria K Shanmugam, Washington D.C., District of Columbia, United States